CLINICAL TRIAL: NCT05758103
Title: Limosilactobacillus Reuteri as an Adjuvant in the Treatment of Peri-implant Mucositis in Total Rehabilitation: an Exploratory Study
Brief Title: Limosilactobacillus Reuteri as an Adjuvant in the Treatment of Peri-implant Mucositis
Acronym: LRRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Malo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LRRCT
Record Dates: First submitted 2023-02-23; First posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Peri-implant Mucositis
Keywords: probiotic; Limosilactobacillus reuteri; dental implant; peri-implant mucositis; total rehabilitation; mechanical therapy; nonsurgical treatment

STUDY DESIGN:
Intervention Model Description: two-group parallel design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mechanical debridement + probiotic supplement (Experimental): Patients with peri-implant mucositis treated through non-surgical professional mechanical debridement and probiotic supplement Limosilactobacillus reuteri Prodentis® (combining L. reuteri DSM 17938 and L. reuteri ATCC PTA 5289 strains).
  Interventions: Dietary Supplement: Limosilactobacillus reuteri Prodentis® (combining L. reuteri DSM 17938 and L. reuteri ATCC PTA 5289 strains)
- Mechanical debridement (No Intervention): Patients with peri-implant mucositis treated through non-surgical professional mechanical debridement alone

INTERVENTIONS:
Dietary Supplement: Limosilactobacillus reuteri Prodentis® (combining L. reuteri DSM 17938 and L. reuteri ATCC PTA 5289 strains) — Non-surgical professional mechanical debridement and probiotic supplement Limosilactobacillus reuteri Prodentis® (combining L. reuteri DSM 17938 and L. reuteri ATCC PTA 5289 strains)
  Arms: Mechanical debridement + probiotic supplement

SUMMARY:
Mechanical debridement is the traditional method for the treatment of peri-implant mucositis and its success depends on the patient's correct oral hygiene. It is believed that probiotics may help by their ability to modulate the oral biofilm, resulting in anti-inflammatory and anti-bacterial plaque action. The aim of this study is to evaluate the adjuvant effect of the probiotic Limosilactobacillus reuteri in the mechanical treatment of peri-implant mucositis. This study aims to include 32 subjects with implant-supported total rehabilitation and peri-implant mucositis, divided into test and control groups, equally subjected to professional mechanical debridement, with the administration of a daily GUM® PerioBalance® lozenge for 30 days added to the test group. Plaque Index, Bleeding Index and probing pocket depth are evaluated before the intervention (baseline) and at 6 and 10 weeks later.

ELIGIBILITY:
Inclusion Criteria:

(i) dental implants placed for at least 12 months according to the All-on-4® concept;

(ii) removal of the dental prosthesis as part of the conventional implant maintenance protocol;

(iii) modified Bleeding Index19 score >0 in at least one implant in the studied rehabilitation;

(iv) implants connected to the prosthesis by means of transepithelial abutments;

(v) if there were natural teeth in opposing arch, they were periodontally healthy or had been treated for periodontitis and were on periodontal support with residual pockets ≤5mm;

(vi) demonstrated previous compliance with oral hygiene appointments; (vii) read and signed the informed consent.

Exclusion Criteria:

(i) Peri-implantitis proven clinically (implant mobility, suppuration and/or pocket depth (PD) ≥5mm) and/or radiographically (bone remodeling greater than 2mm in the first year of function20 and mean marginal bone loss greater than 0.2mm for each subsequent year21 in the rehabilitated arch that was intended to be studied);

(ii) clinically active peri-implantitis (mobility, suppuration and/or PD ≥5mm) in the opposing arch to the one intended to be studied;

(iii) presence of an extra-maxillary/zygomatic implant in the rehabilitated arch that was intended to be studied;

(iv) current probiotic supplementation;

(v) diabetes mellitus not controlled by medication;

(vi) current use of oral hygiene products containing chlorohexidine or essential oils;

(vii) special needs individuals who depended on others for their oral hygiene and medication uptake.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-09-18 (Actual)

PRIMARY OUTCOMES:
Modified bleeding index | baseline, 6 weeks, 10 weeks
  Change of the bleeding score on each dental implant from baseline to 6 weeks and from baseline to10 weeks.
  Modified bleeding index- 0: absence of bleeding; 1: isolated bleeding spots visible; 2: blood forms a confluent red line on margin; 3: heavy or profuse bleeding.

SECONDARY OUTCOMES:
Modified plaque index | baseline, 6 weeks, 10 weeks
  Change of the bacterial plaque score on each dental implant from baseline to 6 weeks and from baseline to10 weeks.
  Modified plaque index- 0: absence of plaque; 1: plaque only visible after running the periodontal probe through the peri-implant sulcus around the implant; 2: plaque visible by the naked eye; 3: abundance of soft matter.
Probing pocket depth | baseline, 6 weeks, 10 weeks
  Change of the probing pocket depth in milimeters on each dental implant from baseline to 6 weeks and from baseline to10 weeks. Values over 4 mm might indicate the presence of an acute or chronical peri-implant condition.

CONTACTS AND LOCATIONS:
Overall Officials: Gonçalo Parreira, MSc, Principal Investigator — Maló Clinic
Locations (1):
- Malo Clinic, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request to the Principal Investigator
Supporting Information: Study Protocol, SAP